CLINICAL TRIAL: NCT02817763
Title: Evaluation of a New Surgical-restorative Approach for the Treatment of Gingival Recessions Associated With Non-carious Cervical Lesions: a Randomized Controlled Clinical Trial
Brief Title: A New Surgical-restorative Approach to Treat Gingival Recessions Associated With Non-carious Cervical Lesions (NCCL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF 4
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Gingival Recession; Tooth Abrasion
MeSH Terms: conditions — Gingival Recession; Tooth Abrasion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connective tissue graft (CTG) (Active Comparator): After local anesthesia, the surgical procedure performed was the trapezoidal-type of Coronally advanced flap (CAF). After the flap was raised, the exposed root surface was gently scaled and planed until it became smooth. Afterward, a thin and small connective tissue graft that was sutured over the root surface. Then, the flap was coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: Connective tissue graft (CTG); Drug: sodium dipyrone
- CTG plus resin composite restoration (Experimental): After local anesthesia, a sterile rubber dam was placed to isolate the operative field and the coronal zone of the non-carious cervical lesion restoration was performed with a nanocomposite resin, following the manufacturer's instructions. The apical margin of the restoration was place 1 millimeter beyond to the cemento-enamel junction estimation. In the next session, the surgical procedure performed was the trapezoidal-type of CAF. After the trapezoidal-type of CAF flap was raised, a thin and small connective tissue graft that was sutured over the restoration surface. Then, the flap was coronally positioned and sutured to completely cover the graft.
  Interventions: Procedure: CTG plus resin composite restoration; Drug: sodium dipyrone

INTERVENTIONS:
Procedure: Connective tissue graft (CTG) — Periodontal surgical technique to treat gingival recessions
  Other Names: Periodontal plastic surgery
  Arms: Connective tissue graft (CTG)
Procedure: CTG plus resin composite restoration — Periodontal surgical technique to treat gingival recessions Procedure/Surgery: Resin composite restoration Restorative procedure do treat tooth structure loss
  Other Names: Periodontal plastic surgery
  Arms: CTG plus resin composite restoration
Drug: sodium dipyrone — sodium dipyrone was recommended for all participants after the surgical procedures.

SUMMARY:
The aim of the present study is to evaluate the clinical, aesthetic and patient-centered parameters of connective tissue graft associated or not with partial resin composite (RC) for the treatment of gingival recession with NCCL, performed before the surgical procedure.

DETAILED DESCRIPTION:
This was a prospective, parallel and controlled clinical trial.

- Group CTG (control n = 20) - patients who received connective tissue graft to treat gingival recession associated with non-carious cervical lesion. Group CTG+RC (test n = 20) - patients who received connective tissue graft plus partial resin composite restoration to treat gingival recession associated with non-carious cervical lesion.

The surgeries, as well as all postoperative follow-up, were performed at the dental clinic of Institute of Science and Technology (ICT), State University of São Paulo (UNESP). For those recessions allocated to CTG group, two horizontal incisions were made at right angles to the adjacent interdental papillae, without interfering with the gingival margins of neighboring teeth. Two oblique vertical incisions were extended beyond the mucogingival junction, and a trapezoidal mucoperiosteal flap was raised up to the mucogingival junction. After this point, a split-thickness flap was extended apically, releasing the tension and favoring coronal positioning of the flap.The exposed root surface was gently scaled and planed until it became smooth in the CTG group. Afterwards, a thin and small connective tissue graft was removed from the palatal site and sutured over the root surface. Then, the flap was coronally positioned and sutured to completely cover the graft. For those recessions allocated to CTG+RC group, firstly a sterile rubber dam was placed to isolate the operative field and the coronal zone of the non-carious cervical lesion restoration was performed with a nanocomposite resin, following the manufacturer's instructions. The apical margin of the restoration was place 1 millimeter apically to the cemento-enamel junction estimation. In the following session the CTG+RC received the surgical procedure as described above where a thin and small connective tissue graft was removed from the palatal site and sutured over the root/restoration surface. Then, the flap was coronally positioned and sutured to completely cover the graft.

Clinical parameters were assessed at baseline and 3 and 6 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* presenting Miller class I or II gingival recession in the maxillary canines or premolars associated with non-carious cervical lesion;
* teeth included in the study should present pulp vitality;
* patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤ 20%;
* patients older than 18 years old;
* probing depth ˂ 3 mm in the included teeth;
* patients who agreed to participate and signed an informed consent form

Exclusion Criteria:

* patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure
* patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure
* smokers or pregnant women
* patients who underwent periodontal surgery in the area of interest.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santamaria MP, da Silva Feitosa D, Casati MZ, Nociti FH Jr, Sallum AW, Sallum EA. Randomized controlled clinical trial evaluating connective tissue graft plus resin-modified glass ionomer restoration for the treatment of gingival recession associated with non-carious cervical lesion: 2-year follow-up. J Periodontol. 2013 Sep;84(9):e1-8. doi: 10.1902/jop.2013.120447. Epub 2013 Jan 31. PMID 23368948
- [Background] Santamaria MP, Ambrosano GM, Casati MZ, Nociti Junior FH, Sallum AW, Sallum EA. Connective tissue graft plus resin-modified glass ionomer restoration for the treatment of gingival recession associated with non-carious cervical lesion: a randomized-controlled clinical trial. J Clin Periodontol. 2009 Sep;36(9):791-8. doi: 10.1111/j.1600-051X.2009.01441.x. Epub 2009 Jul 7. PMID 19594663
- [Background] Zucchelli G, Gori G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, De Sanctis M. Non-carious cervical lesions associated with gingival recessions: a decision-making process. J Periodontol. 2011 Dec;82(12):1713-24. doi: 10.1902/jop.2011.110080. Epub 2011 May 4. PMID 21542735
- [Derived] Santamaria MP, Silveira CA, Mathias IF, Neves FLDS, Dos Santos LM, Jardini MAN, Tatakis DN, Sallum EA, Bresciani E. Treatment of single maxillary gingival recession associated with non-carious cervical lesion: Randomized clinical trial comparing connective tissue graft alone to graft plus partial restoration. J Clin Periodontol. 2018 Aug;45(8):968-976. doi: 10.1111/jcpe.12907. Epub 2018 Jun 25. PMID 29681059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Pre-assignment Details: The study recruited 45 eligible patients. However, five patients were excluded before assignment to groups. One recruited patient never presented for treatment and four declined to proceed.
Period: Overall Study
Arm/Group | Connective Tissue Graft (CTG) | CTG Plus Resin Composite Restoration
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Connective Tissue Graft (CTG) | CTG Plus Resin Composite Restoration | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.52 (10.26) | 44.35 (10.39) | 44.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 20 | 20 | 40
Gingival recession depth [Mean (Standard Deviation); unit: millimeters] | 3.34 (0.7) | 3.29 (1.13) | 3.31 (0.03)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Defect Coverage
Description: Percentage mean (%) of root surface covered by the surgical treatment, measured through a periodontal probe.
Time Frame: 6 months
Measure: Count of Units; unit: Gingival recessions
Units Other Than Participants: Gingival recessions
Arm/Group | Connective Tissue Graft (CTG) | CTG Plus Resin Composite Restoration
Number analyzed (Participants) | 20 | 20
Number analyzed (Gingival recessions) | 20 | 20
Gingival recessions | 15 | 14

2. Secondary Outcome: Modified Root Coverage Esthetic Score (MRES)
Description: The MRES evaluated six variables: gingival margin (GM): 0 or 3 points; marginal tissue contour (MTC): 0 or 1 point; soft tissue texture (STT): 0 or 1 point; mucogingival junction alignment (MGJ): 0 or 1 point; gingival color (GC): 0 or 1 point; restoration/cervical lesion color (R/CLC): 0 points = color of restoration or uncovered cervical lesion does not match with tooth's color; 3 points = good color integration. Thus, 10 points was a perfect score.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: photographs
Arm/Group | Connective Tissue Graft (CTG) | CTG Plus Resin Composite Restoration
Number analyzed (Participants) | 20 | 20
Number analyzed (photographs) | 40 | 40
units on a scale | 7.13 (0.07) | 8.71 (0.89)

ADVERSE EVENTS:
Arm/Group | Connective Tissue Graft (CTG) | CTG Plus Resin Composite Restoration
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No